CLINICAL TRIAL: NCT04151797
Title: Impact of a Mobile Geriatric Team With a Pharmacist on the Optimisation of Prescriptions in Elderly Inpatients
Acronym: PHARMOG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: RC31/17/0353
Record Dates: First submitted 2019-10-15; First posted 2019-11-05 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2021-05

CONDITIONS: Medication Therapy Management
Keywords: Medication review; clinical pharmacy; polypharmacy; older people; collaboration; inappropriate prescribing
MeSH Terms: interventions — Medication Therapy Management

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Medication therapy management (Experimental): Medication therapy management by pharmacist-led medication review
  Interventions: Other: Medication therapy management

INTERVENTIONS:
Other: Medication therapy management — The intervention is in the form of a pharmacist-led medication review aimed at detecting potentially inappropriate prescribing. It includes:
  * Data collection on comorbidities, medication and laboratory results.
  * A pharmacist's evaluation of the prescriptions based on the patient's conditions and on the current recommendations for clinical practice.
  * A detailed feedback to the geriatrician.
  * A written report addressed to the attending physician

SUMMARY:
In patients aged 75 years and older, polypathology is frequent and often associated with polypharmacy. This polypharmacy coupled with a lack of proactive elderly care can sometimes lead to hospitalisation. Due to comorbidities and complex problems, management of geriatric patients usually requires a multidisciplinary approach. In Toulouse University Hospital, elderly inpatients can benefit from a geriatric assessment by a Geriatric Mobile Team. Whether this team improve the prescriptions through the advice of a clinical pharmacist has not been demonstrated yet.

DETAILED DESCRIPTION:
All participants will be identified via the geriatrician of the mobile geriatric team with the following inclusion criteria: age ≥ 75 years, ≥ 5 medications per day and being hospitalised either in emergency room, short-stay medicine unit or in a surgery department. For each patient, the pharmacist will detect potentially inappropriate prescribing (based on explicit criteria and an implicit approach) and liaise with the geriatrician for drug optimisations. The pharmaceutical advice will be added to the geriatrician's written report, and then addressed to the relevant physician. The implementation of the proposals will be evaluated immediately at the end of hospitalisation, and then reassessed three months later by calling the patient and/or his community pharmacist. A total of 250 patients will be enrolled over a 12 month-period. The evolution of potentially inappropriate prescribing will be assessed and their cost evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 75 or older
* Having 5 medications or more per day
* Being hospitalised either in emergency room, short-stay medicine unit or surgery department

Exclusion Criteria:

* Patient refuses to participate
* Patient already included in another study

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 200 (Actual)
Dates: Start 2019-11-19 (Actual); Primary Completion 2021-03-22 (Actual); Study Completion 2021-03-22 (Actual)

PRIMARY OUTCOMES:
Change from baseline patients' number of potentially inappropriate prescription at the patient discharge after optimization by a mobile geriatric team with pharmacist | Month 0 and max Month 2 (At the patient discharge)
  number of potentially inappropriate prescribing per patient before (month 0) and after the intervention of the mobile geriatric team (at the patient discharge)

SECONDARY OUTCOMES:
Change from baseline patients' number of potentially inappropriate prescription at 3 months after optimization by a mobile geriatric team with pharmacist | Month 0, Month 3
  number of potentially inappropriate prescribing per patient before (month 0) and after the intervention of the mobile geriatric team (month 3)
Change from baseline patients' number with at least one potentially inappropriate drug at 3 months after optimization by a mobile geriatric team with pharmacist | Month 0, Month 3
  number of patients with at least one potentially inappropriate drug before (month 0) and after the intervention of the mobile geriatric team (month 3)
Change from baseline ratio of potentially inappropriate drug per patient at 3 months after optimization by a mobile geriatric team with pharmacist | Month 0, Month 3
  ratio of potentially inappropriate drug per patient before (month 0) and after (month 3) the intervention of the mobile geriatric team.
Change from baseline mean number of medications per patient at 3 months | Month 0, Month 3
  Mean number of medications per patient
realisation of a pharmacist-led medication review in primary care | Month 3
  Number of pharmacist-led medication review performed in primary care at 3 months
number of falls 3 months after pharmacist-led medication review | Month 3
  Number of falls
mortality 3 months after pharmacist-led medication review | Month 3
  Number of deaths
re-hospitalisation, including emergency room transfers | Month 3
  Number of non-scheduled hospitalisations (including emergency department transfers)
The nursing home transfers | Month 3
  Number of nursing home transfers

CONTACTS AND LOCATIONS:
Overall Officials: Philippe CESTAC, PharmD, PhD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- Toulouse University Hospital, Toulouse, Occitanie, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pages A, Roland C, Qassemi S, Abdeljalil AB, Houles M, Romain M, Toulza O, Belloc A, McCambridge C, Voisin T, Cestac P, Juillard-Condat B; PharMoG study group. Impact of a Pharmacist-included Mobile Geriatrics team intervention on potentially inappropriate drug prescribing: protocol for a prospective feasibility study (PharMoG study). BMJ Open. 2020 Dec 2;10(12):e040917. doi: 10.1136/bmjopen-2020-040917. PMID 33268421